CLINICAL TRIAL: NCT06712199
Title: Effect of Oxalidine Combined with Reduced-opioid Anesthesia on Multimodal Analgesia in Morbidly Obese Patients Undergoing Bariatric Surgery: a Prospective, Single-center, Randomized, Parallel Controlled Study
Brief Title: Effect of Oxalidine Combined with Reduced-opioid Anesthesia on Multimodal Analgesia in Morbidly Obese Patients Undergoing Bariatric Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongtao Sun (Other)
Collaborators: The First Hospital affiliated of Shandong First Medical University (Unknown)
Responsible Party: Sponsor-Investigator, Yongtao Sun, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: oxalidine
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Morbid Obesity
Keywords: Oxeridine; Hypopiate anesthesia; Multimodal analgesia; Morbid obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Anesthesia Group (OBA Group) (Placebo Comparator): In OBA group, propofol, rocuronium bromide and sufentanil were induced by combined anesthesia, tracheal intubation was performed through a visual laryngeal mask, propofol and remifentanil were injected into the intraoperative pump to maintain anesthesia, and sufentanil was brided to 10μg 30 minutes before the end of the operation. PCA administration regimen in OBA group: Sufentanil + dexmedetomidine + Ondansetron.
  Interventions: Drug: oxalidine
- Less opioid anesthesia Group (OFA group) (Experimental): In OFA group, propofol, rocuronium bromide and esketamine were induced by combined anesthesia, and endotracheal intubation was performed through visual laryngeal mask. Intraoperative pump propofol and esketamine to maintain anesthesia; Oxeridine was bridged-1.5 mg 30min before the operation and administered in two doses, 0.75mg/ time, with an interval of 10min.
  Interventions: Drug: oxalidine

INTERVENTIONS:
Drug: oxalidine — Opioid anesthesia group (OBA group) Anesthesia was induced with propofol 2.5mg·kg-1, rocuronium 0.6mg·kg-1 and sufentanil 0.3μg·kg-1. When BIS value reached 40-60, tracheal intubation was performed through visual laryngeal mask airway. Anesthesia was maintained with propofol 4-12 mg·kg-1·h-1 and remifentanil 0.2-0.5 μg·kg-1·min-1. Sufentanil 10μg was bridaged 30min before the end of surgery. The PCA dosing regimen was sufentanil 2 µg/kg+ dexmedetomidine 2 µg/kg+ ondansetron 24mg.
  Reduced-opioid anesthesia group (OFA group)
  Anesthesia was induced with propofol 2.5mg·kg-1, rocuronium 0.6mg·kg-1 and esketamine 0.3mg·kg-1. When BIS value reached 40-60, tracheal intubation was performed through visual laryngeal mask airway. Propofol 4-12 mg·kg-1·h-1 and esketamine 0.3-0.5 mg·kg-1·h-1 were pumped to maintain anesthesia during operation. Oxalidine 1.5mg was given in two divided doses of 0.75mg each time with an interval of 10min 30min before the end of surgery. The PCA regimen was as follows:
  Other Names: Less opioids for anesthesia

SUMMARY:
The goal of this study is to elucidate the efficacy and safety of oxelidine combined with oligopiate anesthesia for multi-modal analgesia in weight-loss surgery in morbidly obese patients, and to discover a new strategy for multi-modal analgesia management in weight-loss surgery, laying a foundation for the widespread application of oligopiate anesthesia in special patients.

A total of 124 patients who underwent elective bariatric surgery in our hospital were selected, and the participants were randomly divided into two groups: the opioid anesthesia group (OBA group) and the low-opioid anesthesia group (OFA group) using a random number table to achieve simple randomization.

Inclusion criteria: 1.ASA grade I ~ III; 2. Age ≥18 years old; 3. Bariatric surgery patients with BMI≥35kg/m2 and complex signs of morbid obesity (such as metabolic syndrome) 4. Sign the informed consent form.

Exclusion criteria: 1. Positive pregnancy test or breastfeeding; 2. Patients with a history of substance abuse or dependence on opioids; 3. Patients with chronic pain or with severe heart, lung, liver or nervous system diseases.

Anesthesia implementation: 1. Routine monitoring after entry, intravenous administration of midazolam and atropine. Study participants were placed in the ramp position, bilateral recurrent laryngeal nerve block under ultrasound guidance, and the mouth contained dachronine gel. Radial artery puncture was performed and dexmedetomidine was injected intravenously. A laryngeal tube is used to test the sensation of the back of the oropharynx, and a laryngeal mask is placed while awake to connect the anesthesia circuit and deliver oxygen. Once the vocal cords are seen and the end-respiratory CO2 waveform is observed.

2. The OBA group underwent combined anesthesia induction with propofol, rocuronium bromide and sufentanil, endotracheal intubation through visual laryngeal mask, intraoperative pump injection of propofol and remifentanil to maintain anesthesia, sufentanil bridging 10μg 30 minutes before the end of the operation; In OFA group, propofol, rocuronium bromide and esketamine were induced by combined anesthesia, and endotracheal intubation was performed through visual laryngeal mask. Intraoperative pump propofol and esketamine to maintain anesthesia; Oxeridine was bridged-1.5 mg 30min before the operation and administered in two doses, 0.75mg/ time, with an interval of 10min.

3. Both groups were subjected to bilateral lower costal margin transversal nerve block under ultrasound guidance.

4. Ondansetron was given before the end of the operation. After the operation, the tracheal cannula was removed under deep anesthesia, and the laryngeal mask was retained and transferred to the postoperative resuscitation room. Sugengosaccharide sodium was used to antagonize muscle pine during recovery. After the study participants were awake, the laryngeal mask was well tolerated. The laryngeal mask was removed after observation for 1h, and the laryngeal mask was safely transferred to the ward after continuous observation for 1h.

PCA administration regimen in OBA group: Sufentanil + dexmedetomidine + Ondansetron; OFA group PCA administration regimen: oxelidine + dexmedetomidine + Ondansetron. Record the number of compressions, if the assessment of NRS≥4 points, then remedy 2mg oxycodone hydrochloride, and record the dosage.

Main outcome measures: Consumption of oral morphine equivalent (OME) opioids in the 24 hours prior to surgery.

Secondary outcome measures: Overall satisfaction with analgesia and Numerical Rating Scale (NRS, 0-10) pain score, area under the curve of resting and exercise NRS score (AUC) within 72 hours after surgery, time to first use of rescue analgesics within 72 hours, cumulative opioid consumption 72 hours after surgery (morphine milligram equivalent, morphine milligram equivalent, NRS score) MME), participants' satisfaction with postoperative analgesia, 15-item Quality of Recovery score Scale (QoR15) at 24, 48, and 72h after surgery, incidence of postoperative complications, incidence of nausea and vomiting, and incidence of adverse events were recorded.

DETAILED DESCRIPTION:
In this study, sample size was calculated according to the method of comparing two independent samples from PASS software. A Ahmed SA[1] -based study (an effect of opioid-free anesthesia on postoperative opioid consumption during laparoscopic bariatric surgery: a randomized controlled double-blind study focusing on morphine consumption in the first 24h) was 5.8±1.9mg in the first 24 hours in the OFA group compared with 7.2 ± 2.3 mg in the OBA group. Set bilateral α =0.05, the grasp (1- β) is 90%. The sample size consisted of 49 patients in the OFA group and 49 patients in the control group. Considering 20% loss and refusal, at least 124 cases were included.

This study is a single-center, single-blind, randomized controlled study, select patients undergoing elective weight loss surgery in our hospital, and preoperative screening eligible study participants will voluntarily sign written informed consent before randomization. The study physician is responsible for assigning the interventions. Before the study participants entered the operating room, the special researchers who did not participate in the clinical observation realized the simple randomization method with a random number table. The study participants were randomly divided into two groups. The results were stored in an opaque envelope and not opened until 20 minutes before the start of anesthesia, and the drug extraction and preparation were performed. We selected the same group of surgeons to perform weight-loss surgery for the study participants.

Pre-anesthesia preparation: All study participants considered difficult airway and general anesthesia was placed under a visual laryngeal mask during awake descent. Routine monitored after transport to the operating room, midazolam 2 mg and atropine 0.4 mg were administered intravenously. Study participants placed slope position, ultrasound-guided bilateral recurrent laryngeal nerve block, injected 0.375% ropivacaine 2 mL, 10 mL mouth containing 10min. Monitoring invasive arterial blood pressure under local anesthesia, dexmedetomidine (load amount 1 μ g · kg-1 · 10min-1, maintenance amount 0.5 μ g · kg-1 · h-1 to 40min before the end of surgery). Test the sensation of the back of the oropharynx with a anesthetic tube. If there is a nausea reflex, locally spray 2% lidocaine 2 mL in the back of the oropharynx with a tube. The laryngeal mask model was selected according to the lean body weight of the study participants, and the laryngeal mask was placed in the awake state. All the study participants were well tolerated, connected to the anesthesia circuit, and delivered 100% oxygen. Once the vocal cords are seen, and the terminal respiratory carbon dioxide waveform is observed.

anesthesia induction: Opioid anesthesia group (OBA group): propofol 2.5mg · kg-1, rocuronium and 0.6mg · kg-1 and sufentanil 0.3 μ g · kg-1 combined anesthesia induction, endotracheal intubation through visual laryngeal mask when BIS value reaches 40-60; Less opioid anesthesia group (OFA group): propofol 2.5mg · kg-1, rocuronium and 0.6mg · kg-1 and esketamine 0.3mg · kg-1 combined anesthesia induction, endotracheal intubation through visual laryngeal mask when BIS value reaches 40~60; Participants in both groups retained laryngeal mask evacuated cuff gas and applied endotracheal intubation to maintain anesthesia. Select 0.375% ropivacaine 40 mL, both groups were compound ultrasound guided downward bilateral inferior transverse abdominal muscle nerve block.

continuous anesthesia: Opioid anesthesia group (OBA group): pump propofol 4-12 mg · kg-1 · h-1 and remifentanil 0.2-0.5 μ g · kg-1 · min-1 for maintenance anesthesia; bridge sufentanyl 10 μ g 30min before surgery.

Less-opioid anesthesia group (OFA group): pump propofol 4-12 mg · kg-1 · h-1 and esketamine 0.3~0.5mg · kg-1 · h-1 maintenance anesthesia; bridging oslilidine 1.5mg 30min before surgery, 0.75mg / dose, 10min interval.

Both groups were ventilated with tidal volume of 6 ~ 8 mL/Kg to avoid barotrauma, respiratory rate 10~14 breaths / min, positive end-expiratory pressure (PEEP) 5~10 cmH2O to maintain PETCO2 35~45 cmH2O. We considered hemodynamic instability as SAE (vasoactive drugs for hypotension or hypertension, atropine for bradycardia, β blockers for tachycardia) and recorded the number of treatments. Ondansetron (8mg, iv) was given 20 min before the end of the operation. After surgery, the endotracheal intubation was removed under deep anesthesia, and the laryngeal mask was retained and transferred to the postoperative resuscitation room (PACU). During the resuscitation period, 2 to 4 mg · kg-1. After the study participants were awake, the laryngeal mask was well tolerated, and the laryngeal mask was removed 1h after observation and safely transferred to the ward after further observation for 1h.

Postoperative pain management:

PCA dosing regimen in the opioid anesthesia group (OBA group): sufentanyl 2 µ g / kg + dexmedetomidine 2 µ g / kg + ondansetron 24mg; PCA dosing regimen in the less-opioid anesthesia group (OFA group): Osiidine 30mg + dexmedetomidine 2 µ g / kg + ondansetron 24mg.

Both groups were configured to 100ml, with a background dose of 2ml / h, a bolus volume of 0.5ml / time, and a locking time of 15min. Record the number of presses, if you evaluate the NRS 4 points, remedy oxycodone hydrochloride 2mg, and record the dosage.

Study intervention program Opioid Anesthesia Group (OBA group) Propofol 2.5mg · kg-1, rocuronium and 0.6mg · kg-1 and sufentanil 0.3 μ g · kg-1 for BIS at 40-60; pump propofol 4-12 mg · kg-1 · h-1 and remifentanil 0.2~0.5 μ g · kg-1 · min-1 to maintain anesthesia; 10 μ g 30min before surgery. PCA dosing regimen: sufentanyl 2 µ g / kg + dexmedetomidine 2 µ g / kg + ondansetron 24mg.

Less-opioid anesthesia group (OFA group) Propofol 2.5mg · kg-1, rocuronium and 0.6mg · kg-1 and esketamine 0.3mg · kg-1 combined anesthesia induction, tracheal intubation at 40-60; pump propofol 4-12 mg · kg-1 · h-1 and esketamine 0.3~0.5mg · kg-1 · h-1; maintain anesthesia, bridging Osilidine 1.5mg 30min before surgery, administered twice, 0.75mg / time, 10min interval. PCA dosing regimen: Oliidine 30mg + dexmedetomidine 2 µ g / kg + ondansetron 24mg.

Determination of analgesic effect and analgesic remedial measures During hospitalization, if NRS score 4,2mg for rescue analgesia; if score 7 exceeds 24h, this will be defined as an adverse event and all details will be recorded in the CRF.

Recording and handling of adverse events Pain: If the NRS score is ≥4, 2mg oxycodone should be injected intravenously for rescue and analgesia.

Agitation: The assessment was made using the Richmond Agitation sedation Score (RASS). If the score was ≥+2, sedation was given (dexmedetomine drops were given according to body weight).

Delirium: The 3D-CAM delirium scale was used to assess, and if delirium occurred, sedation was administered (dexmetopidine intravenous drops according to body weight); Respiratory depression: defined as SpO2 < 90%, if respiratory depression occurs, immediately adjust the oxygen flow, mask pressure ventilation if necessary; Respiratory depression should be monitored during anesthesia induction and recovery to ensure the safety of study participants.

Delayed recovery: defined as residual sedation for more than 30 minutes after withdrawal, where appropriate, flumaxinil antagonism is given; Postoperative chills: Wrench standard grading: 0, no chills; Grade 1, fasciculus and/or peripheral vascular constriction and/or peripheral cyanosis, but no muscle fibrillation; Grade 2, only one muscle group fibrillation; Grade 3, more than one muscle group muscle fibrillation; Level 4, generalized fibrillation. Wrench score ≥3 is defined as the occurrence of chills. If study participants developed chills, they were treated with pethidine hydrochloride injection; Postoperative nausea and vomiting: PONV was assessed using grades (grade 1: mild nausea, abdominal discomfort, but no vomiting; Grade 2: transient vomiting, vomiting ≤1 time; Grade 3: Vomiting requiring medical treatment, vomiting ≤2 times; Grade 4: Medically difficult to control vomiting, vomiting ≥3 times.) 4.3.6.8 Fluctuations in Blood pressure: When systolic blood pressure (SBP) drops by more than 20% of the baseline value or less than 90mmHg, norepinephrine is given 4μg; When the increase of SBP was more than 20% of the basic value or more than 180mmHg, urapidil 12.5-25 mg was given; 4.3.6.9 Heart rate change: Atropine was given 0.3 ~ 0.5mg when HR < 50 times/hour; HR > 100 times/hour, Esmolol 0.5mg/kg, can be repeated if necessary.

4.3.6.10 Oxelidine overdose or intoxication: presentation of pinpoint pupil, respiratory depression or hypotension. Rescue methods first keep the airway unobstructed, and then give the corresponding support therapy, improve ventilation, oxygen and so on. The relief drug is naloxone, 0.4mg-0.8mg, intravenous injection, necessary time interval 2-3min repeated administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing weight loss surgery under general anesthesia;
* Age ≥18 years old;
* American Society of Anesthesiologists ASA Grade I-III;
* BMI≥35kg/m2 with complex signs of morbid obesity (such as metabolic syndrome)

Exclusion Criteria:

* Pregnancy test positive or breastfeeding;
* Patients with a history of substance abuse or dependence on opioids;
* Patients with chronic pain or with severe heart, lung, liver or nervous system diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral morphine equivalent (OME) opioid consumption in the 24 hours prior to surgery | 24 hours after surgery

SECONDARY OUTCOMES:
Area under the NRS score curve at rest and exercise 72 hours after surgery (AUC) | Within 72 hours after surgery
  Area under the NRS score curve at rest and exercise 72 hours after surgery (AUC)

OTHER OUTCOMES:
Overall satisfaction with analgesia and Numerical Rating Scale (NRS, 0-10) pain scores, study participants' satisfaction with postoperative analgesia, 15-item Quality of Recovery score Scale (QoR15) at 24, 48, and 72h after surgery | 72 hours after surgery
  Numeric Rating Scale (NRS) pain score was used to evaluate the degree of pain. According to the degree of self-rating on a 10-point scale, a total of 1-10 points, according to the corresponding numbers can be divided into different degrees of pain, that is, 0 is no pain, 1 to 3 is mild pain, 4 to 6 is moderate pain, 7 to 10 is severe pain.
  study participants' satisfaction with postoperative analgesia, The QoR-15 scale, which ranges from 0 (very poor quality of recovery) to 150 (excellent quality of recovery), can visually reflect the postoperative recovery status of patients. In addition, the scale has high reliability and validity, and the assessment time is relatively short, usually 3-4 minutes, which facilitates its wide application in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided